CLINICAL TRIAL: NCT04927741
Title: The Use of Topically Applied Sweet Marjoram Essential Oil for Pain Reduction Following IUD Placement
Brief Title: Essential Oils Following IUD Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: IRB00104768; 20-221E (19-812) (Other: Advocate Aurora Research Institute)
Record Dates: First submitted 2021-06-03; First posted 2021-06-16 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Pain, Muscle; IUD
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Intervention Model Description: 1:1:1 Randomization
Who Masked: Participant
Masking Description: Participant will remain blinded until completion of their study activities
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Method 1: Sweet Marjoram Essential Oil + Grapeseed Oil with Massage (Experimental): Subjects randomized will receive dilution of sweet marjoram essential oil (mixed with grapeseed oil), which will be applied topically with massage after IUD insertion.
  Interventions: Other: Sweet Marjoram Essential Oil
- Method 2: Grapeseed Oil with Massage (Active Comparator): Subjects randomized will grapeseed oil applied topically with massage after IUD insertion.
  Interventions: Other: Grapeseed Oil
- Method 3: Control Group (no oil or massage) (No Intervention): Subjects will serve as control and no essential oils or massage will be applied.

INTERVENTIONS:
Other: Sweet Marjoram Essential Oil — Subjects will receive a dilution of sweet marjoram essential oil (15 cc of grapeseed oil with 10 drops of sweet marjoram essential oil).
  Oil will be applied topically by the study medical providers. Providers will wear exam gloves, dip three fingers into the oil solution and apply it topically to the subject's lower abdomen. This will be applied by going left to right for 20 seconds while applying gentle pressure - counter pressure may be applied on the uterus to help relieve cramping.
  Arms: Method 1: Sweet Marjoram Essential Oil + Grapeseed Oil with Massage
Other: Grapeseed Oil — Subjects will receive 15 cc of undiluted grapeseed oil.
  Oil will be applied topically by the study medical providers. Providers will wear exam gloves, dip three fingers into the oil solution and apply it topically to the subject's lower abdomen. This will be applied by going left to right for 20 seconds while applying gentle pressure - counter pressure may be applied on the uterus to help relieve cramping.
  Arms: Method 2: Grapeseed Oil with Massage

SUMMARY:
This study will measure the effects of topical application of sweet marjoram essential oil + grapeseed oil with massage on uterine cramping/pain post-IUD insertion/placement.

The intention is to conduct a pilot study that could give a first look at the data to determine whether this line of research is worth pursuing with more time, effort, and resources. The results of this pilot study will provide adequate data (e.g., variance estimates) needed for obtaining reasonably reliable sample size estimates if larger studies are warranted in the future.

DETAILED DESCRIPTION:
Patients will be consented and randomized to one of three methods by a member of the study team on the day of their IUD insertion. Several variables of interest will be collected via the electronic medical record and via questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of IUD insertion
* English speaking
* Subject has signed study-specific consent form
* Subject has taken clinic recommended NSAID at least 30 minutes prior to IUD insertion

Exclusion Criteria:

* Subject is in post-partum period
* Known allergies to sweet marjoram essential oil or grapeseed oil
* Broken or irritated skin on lower abdomen
* Diagnosis of IBS/IBD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females presenting for IUD placement
Enrollment: 60 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Change in Pain/Discomfort as Assessed by NRS | 15 minutes post oil application/massage
  Pain/discomfort rating change following topical application of sweet marjoram + grapeseed oil with massage after IUD insertion. (Pain/discomfort assessed by NRS on scale of 0-10).

SECONDARY OUTCOMES:
NRS Patient Pain Rating | Within the 15 minutes following oil application/massage
  The secondary objective of this study is to determine ≥ 0.5-point different in perceived pain rating (on a scale of 0-10) exists between Method 1 (sweet marjoram essential oil + grapeseed oil with massage), Method 2 (grapeseed oil with massage), and Method 3 (control group - no oil or massage).

CONTACTS AND LOCATIONS:
Overall Officials: Vicki F Fresen, RNC, MSN, APNP, Principal Investigator — Aurora BayCare Medical Center
Locations (1):
- Aurora BayCare Medical Center, Green Bay, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No